CLINICAL TRIAL: NCT05775289
Title: A Phase II, Randomized, Multicenter, Double-Blind, Controlled Study of Tobemstomig Plus Platinum-Based Chemotherapy Versus Pembrolizumab Plus Platinum-Based Chemotherapy in Patients With Previously Untreated Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study of Tobemstomig Plus Platinum-Based Chemotherapy vs Pembrolizumab Plus Platinum-Based Chemotherapy in Participants With Previously Untreated Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BO44178
Record Dates: First submitted 2023-03-06; First posted 2023-03-20 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Paclitaxel; Pemetrexed; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Tobemstomig + Platinum-Based Chemotherapy (Experimental): Participants with non-squamous (NSQ) NSCLC will receive induction treatment with blinded tobemstomig in combination with pemetrexed and carboplatin, all on Day 1 every 3 weeks (Q3W) for four 21-day cycles, followed by Q3W maintenance therapy with blinded tobemstomig together with pemetrexed until disease progression or treatment discontinuation.
  Participants with squamous (SQ) NSCLC will receive blinded tobemstomig in combination with paclitaxel and carboplatin, all on Day 1 Q3W for four 21 day cycles, followed by blinded tobemstomig (on Day 1) Q3W until disease progression or treatment discontinuation.
  Interventions: Drug: Tobemstomig; Drug: Paclitaxel; Drug: Pemetrexed; Drug: Carboplatin
- Arm B: Pembrolizumab + Platinum-Based Chemotherapy (Active Comparator): Participants with NSQ NSCLC will receive induction treatment with blinded pembrolizumab in combination with pemetrexed and carboplatin, all on Day 1 Q3W for four 21-day cycles, followed by a maintenance therapy with blinded pembrolizumab together with pemetrexed Q3W until disease progression or treatment discontinuation.
  Participants with SQ NSCLC will receive blinded pembrolizumab in combination with paclitaxel and carboplatin, all on Day 1 Q3W for four 21-day cycles, followed by blinded pembrolizumab (on Day 1) Q3W until disease progression or treatment discontinuation.
  Interventions: Drug: Pembrolizumab; Drug: Paclitaxel; Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: Tobemstomig — Participants will receive intravenous (IV) tobemstomig for four 21-day cycles
  Other Names: RO7247669
  Arms: Arm A: Tobemstomig + Platinum-Based Chemotherapy
Drug: Pembrolizumab — Participants will receive IV pembrolizumab four 21-day cycles
  Arms: Arm B: Pembrolizumab + Platinum-Based Chemotherapy
Drug: Paclitaxel — Participants will receive IV paclitaxel Q3W for four 21-day cycles
Drug: Pemetrexed — Participants will receive IV pemetrexed Q3W until disease progression or unacceptable toxicity
Drug: Carboplatin — Participants will receive IV carboplatin Q3W for four 21-day cycles

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and pharmacokinetics of tobemstomig (RO7247669) in combination with platinum-based chemotherapy compared with pembrolizumab plus platinum-based chemotherapy in participants with previously untreated, locally advanced, unresectable (Stage IIIB/IIIC) or metastatic (Stage IV) non-small-cell lung cancer (NSCLC) who are not eligible to receive curative surgery and/or definitive chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Histologically or cytologically documented locally advanced, unresectable (Stage IIIB/IIIC) or metastatic (Stage IV) NSCLC who are not eligible for curative surgery and/or definitive chemoradiotherapy
* No prior systemic treatment for metastatic NSCLC
* Known tumor PD-L1 status
* Confirmed availability of representative tumor specimens
* Measurable disease
* Life expectancy of at least 12 weeks
* Adequate hematologic and end-organ function
* Negative for HIV, hepatitis B (HBV), and hepatitis C (HCV)
* Adequate cardiovascular function

Exclusion Criteria:

* NSCLC known to have a mutation in the EGFR gene or an ALK fusion oncogene
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* Untreated or clinically unstable spinal cord confession
* History of leptomeningeal disease
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once a month or more frequently)
* Uncontrolled or symptomatic hypercalcemia
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, granulomatosis with polyangiitis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with exceptions defined by the protocol
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on the screening chest computed tomography (CT) scan
* Active tuberculosis (TB) or untreated latent TB
* Current treatment with anti-viral therapy for HBV or HCV
* Significant cardiovascular disease within 3 months prior to randomization
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* History of malignancy other than NSCLC within 5 years prior to randomization, with the exception of malignancies with a negligible risk of metastasis or death e.g., 5-year OS] rate > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal breast carcinoma in situ, or Stage I uterine cancer
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that could affect patient safety
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment
* Prior allogeneic stem cell or solid organ transplantation
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during study treatment or within 5 months after the final dose of study treatment
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Any anti-cancer therapy, including hormonal therapy, within 21 days prior to initiation of study treatment
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including, but not limited to, anti-cytotoxic T lymphocyte-associated protein 4, anti-T cell immunoreceptor with Ig and tyrosine-based inhibition motif domains, anti-PD-1 and anti-PD-L1 therapeutic antibodies, and anti-LAG3) agents
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin-2) within 4 weeks or 5 drug-elimination half lives (whichever is longer) prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies, fusion proteins, or platinum-containing compounds
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the tobemstomig or pembrolizumab formulation
* Known allergy or hypersensitivity or other contraindication to any component of the chemotherapy regimen the patient may receive during the study
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2026-06-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-LaRoche
Locations (50):
- United States (2):
  - Henry Ford Health System, Detroit, Michigan
  - Renown Regional Medical Center Hospital, Reno, Nevada
- Australia (4):
  - Westmead Hospital, Westmead, New South Wales
  - Lyell McEwin Hospital, Adelaide, South Australia
  - Barwon Health, Geelong, Victoria
  - Monash Health, Melbourne, Victoria
- Belgium (4):
  - UZ Brussel, Brussels
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - UZ Leuven Gasthuisberg, Leuven
  - AZ St Maarten Campus Leopoldstr, Mechelen
- Brazil (6):
  - Crio - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Nucleo de Oncologia da Bahia - NOB, Salvador, Bahia, Estado de Bahia
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre X, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
- France (4):
  - Centre Leon Berard, Lyon
  - Hopital Cochin, Paris
  - Ico Rene Gauducheau, Saint-Herblain
  - CHU de Toulouse - Hôpital Larrey, Toulouse
- Germany (5):
  - Uniklinik Essen, Essen
  - LungenClinic Großhansdorf GmbH, Großhansdorf
  - Krankenhaus Martha-Maria Halle-Doelau, Halle
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - Lungenfachklinik Immenhausen, Immenhausen
- Italy (7):
  - Azienda Ospedaliera San Giuseppe Moscati, Avellino, Campania
  - AZ.Osp S. Orsola ? Malpighi-Reparto di Oncologia Medica, Bologna, Emilia-Romagna
  - Policlinico Universitario "Agostino Gemelli", Rome, Lazio
  - IRCCS AOU San Martino - IST, Genoa, Liguria
  - Irccs Istituto Europeo di Oncologia (IEO), Milan, Lombardy
  - Asst Di Monza, Monza, Lombardy
  - IOV - Istituto Oncologico Veneto - IRCCS, Padua, Veneto
- Mexico (3):
  - ONCARE Viaducto Napoles, Mexico City, Mexico CITY (federal District)
  - AMIISTO Atencion Medica Integral Investigacion y Terapia Oncologica S.A de C.V, Mexico City, Mexico CITY (federal District)
  - Instituto Nacional de Cancerologia, Distrito Federal
- South Korea (4):
  - Pusan National University Hospital, Busan
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (6):
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Institut Catala d Oncologia Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña, LA Coruna
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
- Turkey (Türkiye) (5):
  - Memorial Ankara Hastanesi, Ankara
  - Ankara City Hospital, Ankara
  - Trakya Universitesi Tip Fakultesi, Medikal Onkoloji Bilim Dali, Balkan Yerleskesi, Edirne
  - Medipol University Medical Faculty, Istanbul
  - ?zmir Medical Park, Izm?r

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female participants ages at least 18 years with previously untreated locally advanced or metastatic non-small cell lung cancer.
Groups:
- Pembro + Chemotherapy (Squamous): Participants with squamous non small-cell lung cancer (NSCLC) received blinded pembrolizumab (pembro) in combination with paclitaxel and carboplatin on Day 1 every three weeks (Q3W) for four 21-day cycles, followed by blinded pembro with pemetrexed Q3W until disease progression or treatment discontinuation for a maximum of 24 months of treatment.
- Pembro + Chemotherapy (Non-squamous): Participants with non-squamous (NSQ) NSCLC received induction treatment with blinded pembro in combination with pemetrexed and carboplatin on Day 1 Q3W for four 21-day cycles, followed by maintenance therapy with blinded pembro with pemetrexed Q3W until disease progression or treatment discontinuation for a maximum of 24 months of treatment.
- Tobe + Chemotherapy (Squamous): Participants with SQ NSCLC received blinded tobemstomig in combination with paclitaxel and carboplatin on Day 1 Q3W until disease progression or treatment discontinuation for a maximum of 24 months of treatment.
- Tobe + Chemotherapy (Non-squamous): Participants with NSQ NSCLC received induction treatment with blinded tobemstomig in combination with pemetrexed and carboplatin on Day 1 Q3W for four 21-day cycles, followed by Q3W maintenance therapy with blinded tobemstomig with pemetrexed until disease progression or treatment discontinuation for a maximum of 24 months of treatment.
Period: Overall Study
Arm/Group | Pembro + Chemotherapy (Squamous) | Pembro + Chemotherapy (Non-squamous) | Tobe + Chemotherapy (Squamous) | Tobe + Chemotherapy (Non-squamous)
Started | 25 | 66 | 24 | 67
Completed | 0 | 0 | 0 | 0
Not Completed | 25 | 66 | 24 | 67
Not completed — Study Ongoing | 20 | 53 | 15 | 55
Not completed — Death | 4 | 11 | 8 | 12
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pembro + Chemotherapy (Non-squamous): Participants with non-squamous NSCLC received induction treatment with blinded pembro in combination with pemetrexed and carboplatin on Day 1 Q3W for four 21-day cycles, followed by maintenance therapy with blinded pembro with pemetrexed Q3W until disease progression or treatment discontinuation for a maximum of 24 months of treatment.
- Total: Total of all reporting groups
Arm/Group | Pembro + Chemotherapy (Squamous) | Pembro + Chemotherapy (Non-squamous) | Tobe + Chemotherapy (Squamous) | Tobe + Chemotherapy (Non-squamous) | Total
Number analyzed (Participants) | 25 | 66 | 24 | 67 | 182
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.2 (6.8) | 63.2 (9.6) | 63.0 (11.2) | 64.8 (8.3) | 64.2 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 27 | 8 | 24 | 64
  Male | 20 | 39 | 16 | 43 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 10 | 5 | 7 | 29
  Not Hispanic or Latino | 18 | 49 | 17 | 53 | 137
  Unknown or Not Reported | 0 | 7 | 2 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 0 | 3
  Asian | 4 | 10 | 3 | 5 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 5 | 0 | 0 | 5
  White | 18 | 40 | 19 | 53 | 130
  More than one race | 0 | 0 | 0 | 2 | 2
  Unknown or Not Reported | 2 | 10 | 1 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from randomization to the first occurrence of disease progression or death from any cause (whichever occurs first), as determined by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Time Frame: Randomization to date of first documented disease progression or death (up to approximately 15 months)
Population: The analysis population included all participants that were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Pembro + Chemotherapy: Participants with squamous or non-squamous NSCLC received induction treatment with blinded pembro in combination with pemetrexed and carboplatin on Day 1 Q3W for four 21-day cycles, followed by maintenance therapy with blinded pembro with pemetrexed Q3W until disease progression or treatment discontinuation for a maximum of 24 months of treatment.
- Tobe + Chemotherapy: Participants with squamous or NSQ NSCLC received induction treatment with blinded tobemstomig in combination with pemetrexed and carboplatin on Day 1 Q3W for four 21-day cycles, followed by Q3W maintenance therapy with blinded tobemstomig with pemetrexed until disease progression or treatment discontinuation for a maximum of 24 months of treatment.
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 91 | 90
Months | 7.13 [5.59 to NA] — Value is NA due to insufficient number of participants with the event. | 7.62 [5.62 to NA] — Value is NA due to insufficient number of participants with the event.
Statistical Analysis 1: Comparison: Pembro + Chemotherapy vs Tobe + Chemotherapy; Test type: Superiority; p = 0.9705, Log Rank; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.63 to 1.56]

2. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants who experience a complete reponse or partial response on two consecutive occasions at least 4 weeks apart as determined by the investigator according to RECIST v1.1.
Time Frame: Up to approximately 15 months
Population: The analysis population was all randomized participants with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 91 | 90
Percent of participants | 46.2 [36.28 to 56.34] | 41.1 [31.51 to 51.44]
Statistical Analysis 1: Comparison: Pembro + Chemotherapy vs Tobe + Chemotherapy; Test type: Superiority; p = 0.4056, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.42 to 1.43]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to death from any cause.
Time Frame: From randomization to death from any cause (up to approximately 15 months)
Population: The efficacy analysis population consisted of all participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 91 | 90
Months | NA [13.37 to NA] — Value is NA due to insufficient number of participants with the event. | 13.17 [12.02 to NA] — Value is NA due to insufficient number of participants with the event.

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first.
Time Frame: From the first occurrence of a confirmed objective response to disease progression or death from any cause (whichever occurs first) (up to approximately 15 months)
Population: The DOR analysis population consisted of participants who achieved an objective response to study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 42 | 37
Months | NA [9.7 to NA] — Value is NA due to insufficient number of participants with the event. | NA [NA to NA] — Value is NA due to insufficient number of participants with the event.

5. Secondary Outcome: PFS in Participants With PD-L1 Expression
Time Frame: Up to 28 months
Reporting Status: Not Posted

6. Secondary Outcome: OS for Participants With PD-L1 Expression
Time Frame: Up to 28 months
Reporting Status: Not Posted

7. Secondary Outcome: Change in Participant-reported Outcomes as Assessed by the European Organisation for Research and Treatment (EORTC): Physical Functioning
Description: The EORTC Item Library 17 (IL17) physical functioning scale measures a participant's ability to perform a variety of physical activities. Raw scores are calculated by estimating the average of the items that contribute to the scale. Linear transformation is then used to standardize the raw score to a total score range of 0-100. Higher scores for this measure indicate better outcomes.
Time Frame: Baseline to week 12
Population: The analysis population for patient-reported outcomes (PROs) includes all randomized participants. Baseline PRO measurements were taken prior to Cycle 1 Day 1, resulting in few or no data points for that timepoint.
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 91 | 90
Scores on a scale
  Baseline: number analyzed (Participants) | 86 | 86
  Baseline | 86.67 [6.7 to 100.0] | 80.00 [0.0 to 100.0]
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 1 Day 1 |  | 93.3 [93.3 to 93.3]
  Cycle 2 Day 1: number analyzed (Participants) | 82 | 80
  Cycle 2 Day 1 | 80.00 [20.0 to 100.0] | 80.00 [0.0 to 100.0]
  Cycle 3 Day 1: number analyzed (Participants) | 79 | 73
  Cycle 3 Day 1 | 80.00 [20.0 to 100.0] | 80.00 [20.0 to 100.0]
  Cycle 4 Day 1: number analyzed (Participants) | 75 | 67
  Cycle 4 Day 1 | 86.67 [6.7 to 100.0] | 80.00 [6.7 to 100.0]

8. Secondary Outcome: Change in Participant-reported Outcomes as Assessed by the EORTC: Global Health Status/Quality of Life (GHS/QoL)
Description: The EORTC Item Library 17 (IL17) Global Health Status/Quality of Life (GHS/QoL) scale measures the participant's overall health and quality of health over the last week. Raw scores are calculated by estimating the average of the items that contribute to the scale. Linear transformation is then used to standardize the raw score to a total score range of 0-100. Higher scores for this measure indicate a higher quality of life.
Time Frame: Baseline to week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 91 | 90
Scores on a scale
  Baseline: number analyzed (Participants) | 86 | 86
  Baseline | 66.67 [0.0 to 100.0] | 66.67 [0.0 to 100.0]
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 1 Day 1 |  | 83.3 [83.3 to 83.3]
  Cycle 2 Day 1: number analyzed (Participants) | 82 | 81
  Cycle 2 Day 1 | 66.67 [0.0 to 100.0] | 66.67 [16.7 to 100.0]
  Cycle 3 Day 1: number analyzed (Participants) | 79 | 73
  Cycle 3 Day 1 | 66.67 [0.0 to 100.0] | 66.67 [0.0 to 100.0]
  Cycle 4 Day 1: number analyzed (Participants) | 75 | 67
  Cycle 4 Day 1 | 66.67 [0.0 to 100.0] | 66.67 [0.0 to 100.0]

9. Secondary Outcome: Change in Participant-reported Outcomes as Assessed by the EORTC: Role Functioning
Description: The EORTC Item Library 17 (IL17) role functioning scale measures the degree to which disease or treatment interferes with the participant's work or daily activities. Raw scores are calculated by estimating the average of the items that contribute to the scale. Linear transformation is then used to standardize the raw score to a total score range of 0-100. Higher scores for this measure indicate better outcomes.
Time Frame: Baseline to week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 91 | 90
Scores on a scale
  Baseline: number analyzed (Participants) | 86 | 86
  Baseline | 91.67 [0.0 to 100.0] | 83.33 [0.0 to 100.0]
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 1 Day 1 |  | 83.3 [83.3 to 83.3]
  Cycle 2 Day 1: number analyzed (Participants) | 82 | 81
  Cycle 2 Day 1 | 83.33 [0.0 to 100.0] | 83.33 [0.0 to 100.0]
  Cycle 3 Day 1: number analyzed (Participants) | 79 | 73
  Cycle 3 Day 1 | 66.67 [0.0 to 100.0] | 83.33 [0.0 to 100.0]
  Cycle 4 Day 1: number analyzed (Participants) | 75 | 67
  Cycle 4 Day 1 | 83.33 [0.0 to 100.0] | 83.33 [0.0 to 100.0]

10. Secondary Outcome: Change in Participant-reported Outcomes as Assessed by the EORTC: Lung Cancer Symptoms/How Much Did You Cough
Description: The EORTC IL 85 lung cancer symptoms/how much did you cough measure assesses the severity and frequency of coughing over the past week. The single item is scored on a scale of 1-4, with higher scores indicating worse outcomes.
Time Frame: Baseline to week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 91 | 90
Scores on a scale
  Baseline: number analyzed (Participants) | 86 | 88
  Baseline | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 1 Day 1 |  | 1.00 [1.0 to 1.0]
  Cycle 2 Day 1: number analyzed (Participants) | 82 | 81
  Cycle 2 Day 1 | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]
  Cycle 3 Day 1: number analyzed (Participants) | 78 | 73
  Cycle 3 Day 1 | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]
  Cycle 4 Day 1: number analyzed (Participants) | 75 | 68
  Cycle 4 Day 1 | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]

11. Secondary Outcome: Change in Participant-reported Outcomes as Assessed by the EORTC: Short of Breath When Rested
Description: The EORTC IL 85 short of breath when rested measure assesses the degree of difficulty breathing while resting over the past week. The single item is scored on a scale of 1-4, with higher scores indicating worse outcomes.
Time Frame: Baseline to week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 91 | 90
Scores on a scale
  Baseline: number analyzed (Participants) | 86 | 88
  Baseline | 1.00 [1.0 to 4.0] | 1.00 [1.0 to 4.0]
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 1 Day 1 |  | 1.00 [1.0 to 1.0]
  Cycle 2 Day 1: number analyzed (Participants) | 82 | 81
  Cycle 2 Day 1 | 1.00 [1.0 to 3.0] | 1.00 [1.0 to 4.0]
  Cycle 3 Day 1: number analyzed (Participants) | 78 | 73
  Cycle 3 Day 1 | 1.00 [1.0 to 4.0] | 1.00 [1.0 to 3.0]
  Cycle 4 Day 1: number analyzed (Participants) | 75 | 68
  Cycle 4 Day 1 | 1.00 [1.0 to 4.0] | 1.00 [1.0 to 2.0]

12. Secondary Outcome: Change in Participant-reported Outcomes as Assessed by the EORTC: Short of Breath When Walked
Description: The EORTC IL 85 short of breath when walked measure assesses the degree of difficulty breathing while walking over the past week. The single item is scored on a scale of 1-4, with higher scores indicating worse outcomes.
Time Frame: Baseline to week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 91 | 90
Scores on a scale
  Baseline: number analyzed (Participants) | 85 | 88
  Baseline | 1.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 1 Day 1 |  | 1.00 [1.0 to 1.0]
  Cycle 2 Day 1: number analyzed (Participants) | 81 | 81
  Cycle 2 Day 1 | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]
  Cycle 3 Day 1: number analyzed (Participants) | 77 | 73
  Cycle 3 Day 1 | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]
  Cycle 4 Day 1: number analyzed (Participants) | 75 | 68
  Cycle 4 Day 1 | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]

13. Secondary Outcome: Change in Participant-reported Outcomes as Assessed by the EORTC: Short of Breath Climbed Stairs
Description: The EORTC IL 85 short of breath climbed stairs measure assesses the degree of difficulty breathing while climbing stairs over the past week. The single item is scored on a scale of 1-4, with higher scores indicating worse outcomes.
Time Frame: Baseline to week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 91 | 90
Scores on a scale
  Baseline: number analyzed (Participants) | 86 | 86
  Baseline | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 1 Day 1 |  | 2.00 [2.0 to 2.0]
  Cycle 2 Day 1: number analyzed (Participants) | 81 | 79
  Cycle 2 Day 1 | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]
  Cycle 3 Day 1: number analyzed (Participants) | 77 | 73
  Cycle 3 Day 1 | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]
  Cycle 4 Day 1: number analyzed (Participants) | 75 | 68
  Cycle 4 Day 1 | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]

14. Secondary Outcome: Change in Participant-reported Outcomes as Assessed by the EORTC: Pain in Chest
Description: The EORTC IL 85 pain in chest measure assesses the severity of chest pain over the past week. The single item is scored on a scale of 1-4, with higher scores indicating worse outcomes.
Time Frame: Baseline to week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 91 | 90
Scores on a scale
  Baseline: number analyzed (Participants) | 86 | 88
  Baseline | 1.00 [1.0 to 3.0] | 1.00 [1.0 to 4.0]
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 1 Day 1 |  | 1.00 [1.0 to 1.0]
  Cycle 2 Day 1: number analyzed (Participants) | 82 | 81
  Cycle 2 Day 1 | 1.00 [1.0 to 3.0] | 1.00 [1.0 to 3.0]
  Cycle 3 Day 1: number analyzed (Participants) | 78 | 73
  Cycle 3 Day 1 | 1.00 [1.0 to 3.0] | 1.00 [1.0 to 4.0]
  Cycle 4 Day 1: number analyzed (Participants) | 75 | 68
  Cycle 4 Day 1 | 1.00 [1.0 to 3.0] | 1.00 [1.0 to 3.0]

15. Secondary Outcome: Change in Participant-reported Outcomes as Assessed by the EORTC: Need to Rest
Description: The EORTC IL 132 need to rest measure assesses how often the participant felt the need to rest over the past week. The single item is scored on a scale of 1-4, with higher scores indicating worse outcomes.
Time Frame: Baseline to week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 91 | 90
Scores on a scale
  Baseline: number analyzed (Participants) | 86 | 88
  Baseline | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 1 Day 1 |  | 2.00 [2.0 to 2.0]
  Cycle 2 Day 1: number analyzed (Participants) | 82 | 81
  Cycle 2 Day 1 | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]
  Cycle 3 Day 1: number analyzed (Participants) | 78 | 73
  Cycle 3 Day 1 | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]
  Cycle 4 Day 1: number analyzed (Participants) | 75 | 68
  Cycle 4 Day 1 | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]

16. Secondary Outcome: Change in Participant-reported Outcomes as Assessed by the EORTC: Felt Weak
Description: The EORTC IL 132 felt weak measure assesses how often the participant felt weak over the past week. The single item is scored on a scale of 1-4, with higher scores indicating worse outcomes.
Time Frame: Baseline to week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 91 | 90
Scores on a scale
  Baseline: number analyzed (Participants) | 86 | 88
  Baseline | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 1 Day 1 |  | 2.00 [2.0 to 2.0]
  Cycle 2 Day 1: number analyzed (Participants) | 82 | 81
  Cycle 2 Day 1 | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]
  Cycle 3 Day 1: number analyzed (Participants) | 78 | 73
  Cycle 3 Day 1 | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]
  Cycle 4 Day 1: number analyzed (Participants) | 75 | 68
  Cycle 4 Day 1 | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]

17. Secondary Outcome: Change in Participant-reported Outcomes as Assessed by the EORTC: Tired
Description: The EORTC IL 132 tired measure assesses how often the participant felt tired over the past week. The single item is scored on a scale of 1-4, with higher scores indicating worse outcomes.
Time Frame: Baseline to week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 91 | 90
Scores on a scale
  Baseline: number analyzed (Participants) | 86 | 88
  Baseline | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 1 Day 1 |  | 2.00 [2.0 to 2.0]
  Cycle 2 Day 1: number analyzed (Participants) | 82 | 81
  Cycle 2 Day 1 | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]
  Cycle 3 Day 1: number analyzed (Participants) | 78 | 73
  Cycle 3 Day 1 | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]
  Cycle 4 Day 1: number analyzed (Participants) | 75 | 68
  Cycle 4 Day 1 | 2.00 [1.0 to 4.0] | 2.00 [1.0 to 4.0]

18. Secondary Outcome: Change in Participant-reported Outcomes as Assessed by the EORTC: Aches/Pain in Bones
Description: The EORTC IL 188 aches/pain in bones measure assessesthe severity of bone pain over the past week. The single item is scored on a scale of 1-4, with higher scores indicating worse outcomes.
Time Frame: Baseline to week 12
Population: as for outcome 7
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 91 | 90
Scores on a scale
  Baseline: number analyzed (Participants) | 86 | 88
  Baseline | 1.00 [1.0 to 4.0] | 1.00 [1.0 to 4.0]
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1
  Cycle 1 Day 1 |  | 1.00 [1.0 to 1.0]
  Cycle 2 Day 1: number analyzed (Participants) | 82 | 81
  Cycle 2 Day 1 | 1.00 [1.0 to 4.0] | 1.00 [1.0 to 4.0]
  Cycle 3 Day 1: number analyzed (Participants) | 79 | 73
  Cycle 3 Day 1 | 1.00 [1.0 to 4.0] | 1.00 [1.0 to 4.0]
  Cycle 4 Day 1: number analyzed (Participants) | 75 | 67
  Cycle 4 Day 1 | 1.00 [1.0 to 4.0] | 1.00 [1.0 to 4.0]

19. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Time Frame: From the start of treatment to 90 days after the final dose of treatment (up to 28 months)
Measure: Number; unit: Count of participants
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 91 | 90
Count of participants | 89 | 89

20. Secondary Outcome: Maximum Serum Concentration (Cmax) of Tobemstomig
Time Frame: Up to approximately 15 months
Population: The pharmacokinetic (PK) population consisted of participants who received IV tobemstomig.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 0 | 88
ug/mL
  Tobe + Paclitaxel + Carboplatin: number analyzed (Participants) | 0 | 24
  Tobe + Paclitaxel + Carboplatin |  | 188 (27.3)
  Tobe + Pemetrexed + Carboplatin: number analyzed (Participants) | 0 | 64
  Tobe + Pemetrexed + Carboplatin |  | 191 (43.1)

21. Secondary Outcome: Time of Maximum Concentration (Tmax) of Tobemstomig
Time Frame: Up to approximately 15 months
Population: The pharmacokinetic (PK) population consisted of participants who received IV tobemstomig.
Measure: Median (Full Range); unit: Day
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 0 | 88
Day
  Tobe + Paclitaxel + Carboplatin: number analyzed (Participants) | 0 | 24
  Tobe + Paclitaxel + Carboplatin |  | 0.0649 [0.0208 to 9.13]
  Tobe + Pemetrexed + Carboplatin: number analyzed (Participants) | 0 | 64
  Tobe + Pemetrexed + Carboplatin |  | 0.0646 [0.0521 to 21]

22. Secondary Outcome: Clearance (CL) of Tobemstomig
Time Frame: Up to approximately 15 months
Population: The pharmacokinetic (PK) population consisted of participants who received IV tobemstomig.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/day
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 0 | 56
mL/day
  Tobe + Paclitaxel + Carboplatin: number analyzed (Participants) | 0 | 14
  Tobe + Paclitaxel + Carboplatin |  | 246 (55.6)
  Tobe + Pemetrexed + Carboplatin: number analyzed (Participants) | 0 | 42
  Tobe + Pemetrexed + Carboplatin |  | 231 (34.5)

23. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Tobemstomig
Time Frame: Up to approximately 15 months
Population: The pharmacokinetic (PK) population consisted of participants who received IV tobemstomig.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 0 | 56
Liters
  Tobe + Paclitaxel + Carboplatin: number analyzed (Participants) | 0 | 14
  Tobe + Paclitaxel + Carboplatin |  | 3.65 (40.2)
  Tobe + Pemetrexed + Carboplatin: number analyzed (Participants) | 0 | 42
  Tobe + Pemetrexed + Carboplatin |  | 3.56 (31.6)

24. Secondary Outcome: Area Under the Concentration-time Curve (AUC) of Tobemstomig
Time Frame: Up to approximately 15 months
Population: The pharmacokinetic (PK) population consisted of participants who received IV tobemstomig.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 0 | 88
day*ug/mL
  Tobe + Paclitaxel + Carboplatin: number analyzed (Participants) | 0 | 24
  Tobe + Paclitaxel + Carboplatin |  | 1470 (31.8)
  Tobe + Pemetrexed + Carboplatin: number analyzed (Participants) | 0 | 64
  Tobe + Pemetrexed + Carboplatin |  | 1500 (114.2)

25. Secondary Outcome: Half-life (T1/2) of Tobemstomig
Time Frame: Up to approximately 15 months
Population: The pharmacokinetic (PK) population consisted of participants who received IV tobemstomig.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 0 | 56
Day
  Tobe + Paclitaxel + Carboplatin: number analyzed (Participants) | 0 | 14
  Tobe + Paclitaxel + Carboplatin |  | 8.45 (196.4)
  Tobe + Pemetrexed + Carboplatin: number analyzed (Participants) | 0 | 42
  Tobe + Pemetrexed + Carboplatin |  | 10.4 (83.2)

26. Secondary Outcome: Percentage of Participants With Anti-drug Antibodies (ADAs)
Time Frame: Baseline up to approximately 15 months
Population: The pharmacokinetic (PK) population consisted of participants who received IV tobemstomig.
Measure: Number; unit: Percentage of participants
Arm/Group | Pembro + Chemotherapy | Tobe + Chemotherapy
Number analyzed (Participants) | 0 | 77
Percentage of participants
  Treatment-Emergent |  | 42.9
  Treatment-Induced |  | 42.9

ADVERSE EVENTS:
Time Frame: From the start of treatment to 90 days after the final dose of treatment (up to 28 months)
Arm/Group | Pembro + Chemotherapy (Squamous) | Pembro + Chemotherapy (Non-squamous) | Tobe + Chemotherapy (Squamous) | Tobe + Chemotherapy (Non-squamous)
All-Cause Mortality (participants affected / at risk) | 4/25 | 11/65 | 8/24 | 12/65
Serious Adverse Events (participants affected / at risk) | 10/25 | 26/65 | 14/24 | 35/65
Other Adverse Events (participants affected / at risk) | 25/25 | 63/65 | 24/24 | 63/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembro + Chemotherapy (Squamous) (N=25) | Pembro + Chemotherapy (Non-squamous) (N=65) | Tobe + Chemotherapy (Squamous) (N=24) | Tobe + Chemotherapy (Non-squamous) (N=65)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 2 (2) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (3) | 6 (8) | 3 (3) | 5 (6)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembro + Chemotherapy (Squamous) (N=25) | Pembro + Chemotherapy (Non-squamous) (N=65) | Tobe + Chemotherapy (Squamous) (N=24) | Tobe + Chemotherapy (Non-squamous) (N=65)
Anaemia (Blood and lymphatic system disorders) | 11 (13) | 40 (52) | 6 (8) | 35 (48)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (5) | 0 (0) | 4 (8)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 16 (22) | 4 (5) | 19 (32)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 8 (13) | 2 (3) | 6 (7)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 1 (2) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 4 (4) | 5 (5) | 9 (10)
Hypothyroidism (Endocrine disorders) | 3 (3) | 4 (4) | 3 (3) | 7 (8)
Lacrimation increased (Eye disorders) | 0 (0) | 10 (12) | 0 (0) | 7 (7)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (6) | 0 (0) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (3) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (6) | 18 (23) | 5 (6) | 22 (25)
Diarrhoea (Gastrointestinal disorders) | 4 (7) | 16 (19) | 7 (7) | 16 (22)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (4) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (7) | 24 (37) | 7 (8) | 32 (43)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 6 (6) | 1 (1) | 5 (5)
Vomiting (Gastrointestinal disorders) | 2 (2) | 7 (7) | 1 (1) | 11 (15)
Asthenia (General disorders) | 5 (6) | 20 (31) | 7 (8) | 21 (42)
Chest pain (General disorders) | 1 (1) | 4 (4) | 0 (0) | 2 (2)
Fatigue (General disorders) | 4 (9) | 14 (17) | 5 (7) | 14 (16)
Mucosal inflammation (General disorders) | 3 (3) | 6 (9) | 2 (2) | 5 (8)
Oedema peripheral (General disorders) | 1 (1) | 5 (6) | 1 (2) | 4 (4)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Pyrexia (General disorders) | 4 (4) | 5 (5) | 1 (1) | 6 (8)
Conjunctivitis (Infections and infestations) | 0 (0) | 5 (6) | 0 (0) | 2 (4)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (4) | 3 (4) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 5 (5) | 0 (0) | 3 (3)
Pneumonia (Infections and infestations) | 2 (2) | 4 (4) | 1 (1) | 6 (6)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 0 (0) | 2 (2) | 3 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 4 (4) | 1 (1) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (4) | 6 (10) | 5 (8)
Alanine aminotransferase increased (Investigations) | 0 (0) | 6 (10) | 2 (2) | 13 (20)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 6 (10) | 3 (4) | 10 (14)
Blood bicarbonate decreased (Investigations) | 0 (0) | 2 (3) | 2 (3) | 2 (3)
Blood creatinine increased (Investigations) | 1 (1) | 4 (5) | 1 (1) | 9 (12)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Lymphocyte count decreased (Investigations) | 1 (2) | 3 (9) | 3 (7) | 3 (9)
Neutrophil count decreased (Investigations) | 1 (2) | 5 (11) | 1 (1) | 4 (7)
Platelet count decreased (Investigations) | 1 (1) | 6 (10) | 1 (1) | 8 (13)
Weight decreased (Investigations) | 2 (2) | 6 (6) | 1 (1) | 5 (5)
White blood cell count decreased (Investigations) | 0 (0) | 4 (5) | 3 (3) | 1 (4)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 15 (22) | 5 (7) | 17 (18)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 7 (8) | 2 (2) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3) | 3 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 6 (9) | 4 (4) | 5 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 7 (10) | 2 (2) | 6 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7) | 7 (7) | 5 (6) | 8 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5) | 2 (2) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5) | 2 (2) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 5 (5) | 1 (1) | 5 (5)
Dysgeusia (Nervous system disorders) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 1 (2) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 8 (8) | 2 (2) | 7 (7) | 3 (3)
Neurotoxicity (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 5 (6) | 2 (2) | 2 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | 5 (5) | 11 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 10 (10) | 4 (4) | 9 (11)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 1 (1) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4) | 4 (4) | 3 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (7) | 9 (11) | 5 (5) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 7 (9) | 11 (13) | 5 (6) | 12 (16)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT05775289/Prot_SAP_000.pdf